CLINICAL TRIAL: NCT05431621
Title: Establishment of Molecular Classification Models for Early Diagnosis of Digestive System Cancers
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Xuhui Central Hospital, Shanghai (Other); Changhai Hospital (Other); Hubei Cancer Hospital (Other); Shanghai Public Health Clinical Center (Other Government); Singlera Genomics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019YFC1315802-01
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer; Gastric (Stomach) Cancer; Colorectal Cancer; Hepatocellular Carcinoma
Keywords: ctDNA markers; DNA methylation; DNA fragment feature; miRNA; CTC; Cancer early detection
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Digestive system cancer group: A total of about 1035 cases are expected to be enrolled, including 432 cases in stage I and 603 cases in II-IV.
- Negative group: 985 healthy individuals.
- High risk group: 410 cases with precancerous diseases.

SUMMARY:
This is a single blind, case control, multicenter study jointly developed by Zhongshan Hospital of Fudan University, Shanghai Public Health Clinical Center, Shanghai Xuhui Central Hospital, Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University, and Shanghai Singlera Genomics Company. The enrolled population will include positive group, precancerous lesions and healthy control group, which is expected to enroll 2,430 participants. The primary objective is to establish molecular testing methods for non-invasive screening and early diagnosis of digestive system cancers through ctDNA methylation and mutation, cfDNA and ctDNA fragment size, and end motif based model (for esophageal, gastric, colorectal cancer), and through ctDNA methylation detection, ctDNA low-pass WGS, miRNA7 and CTC detection and analysis technology based model (for hepatocellular carcinoma). The sensitivity and specificity of the models in cancer early detection will be evaluated.

DETAILED DESCRIPTION:
Design of the project: 1) Participants who sign informed consent forms will complete the disease history information collection;2) Collect samples of cancer tissue and corresponding paracancer samples, as well as peripheral blood; 3) Using the MONOD patent detection data of the company's previous research and combining with literature retrieval, to analyze the tissue samples of digestive system cancers to screen the methylation mutation sites;4) ctDNA methylation markers are preliminarily screened by plasma of healthy persons paired with tissues;5) Using the screened blood ctDNA specific methylation markers together with other molecular markers to establish a targeted detection method for early digestive system cancer lesions;6) Retain the most distinguishing targets in the original panel test and establish the second version of the panel;7) Establish and validate predictive models to finalize multitype molecular target detection for peripheral blood DNA;8) Construct statistical learning models based on ctDNA methylation and fragment features, miRNA7™ and CTC, and optimize the models respectively;9) Evaluate the sensitivity and specificity of the models in cancer early detection.

ELIGIBILITY:
Colorectal cancer, Esophageal cancer and Gastric (stomach) cancer Group

Inclusion Criteria:

1. Aged 18 to 80, no gender limitation, no pregnant or breastfeeding for women;
2. Those who can accept gastroscopy and/or total colonoscopy;
3. Newly-diagnosed patients who had not received surgery, radiotherapy, chemotherapy, targeted therapy or other anti-tumor intervention;
4. Stop anticoagulant drugs such as warfarin, aspirin, and bolivir for 1 week, and stop low molecular weight heparin that day;
5. No previous history of other tumor diseases, and no abnormalities in the liver and kidney;
6. No major trauma requiring blood transfusion treatment within one week.

Exclusion Criteria:

1. Previous esophageal cancer, stomach cancer, bowel cancer and gastrointestinal adenoma;
2. Have a history of other cancers;
3. Systemic inflammatory response syndrome;
4. Previously experienced esophageal, gastric or colorectal adenoma removal or tumor resection;
5. Patients with Lynch syndrome in the family;
6. A history of severe cardiovascular disease (e.g., previous myocardial infarction, coronary artery bypass grafting, coronary stenting, congestive heart failure, myocardial infarction within 6 months, or uncontrolled severe hypertension, etc.) who were deemed unsuitable for inclusion by the investigator;
7. Have participated in an "interventional" clinical trial within the past 30 days and have taken the experimental drug;
8. Unsuitable for this trial determined by the researchers;
9. Failure to collect blood on time according to plan;
10. The blood sample does not meet the requirements.

Hepatocellular Carcinoma Group

Inclusion Criteria:

1. Applicable to all enrolled volunteers (1) Aged 18 to 80, no gender limitation, no pregnant or breastfeeding for women; (2) No previous history of malignancy in other sites; (3) To avoid the risk of bleeding caused by taking anticoagulants during sampling, the following provisions shall be made according to different types of samples: stop anticoagulant drugs such as warfarin, aspirin, and bolivir for 1 week, and stop low molecular weight heparin that day; the doctor in charge decides whether to stop anticoagulant drugs before blood draw, according to the specific situation of the volunteers, ; (4) No major trauma requiring blood transfusion treatment within one week;
2. Only for patients with hepatocellular carcinoma (HCC). (1) Diagnosed with stage I-IV hepatocellular carcinoma; (2) Newly-diagnosed patients with liver cancer, who had not received surgery, radiotherapy, chemotherapy, targeted therapy or other anti-tumor intervention;
3. Only for high-risk groups (1) Diagnosis of child-Pugh grade A or B, chronic hepatitis B or cirrhosis; (2) No history of liver cancer or malignancy in other sites;
4. For healthy people only (1) Normal liver function test results on the day of blood collection; (2) No history of hepatitis B, hepatitis C and cirrhosis; (3) No history of liver cancer or malignancy in other sites.

Exclusion Criteria:

1. Patients with liver cancer who have received surgery, radiotherapy, chemotherapy, targeted therapy;
2. Cancer patients except HCC, or patients with liver metastasis;
3. Systemic inflammatory response syndrome;
4. A history of severe cardiovascular disease (e.g., previous myocardial infarction, coronary artery bypass grafting, coronary stenting, congestive heart failure, myocardial infarction within 6 months, or uncontrolled severe hypertension, etc.) who were deemed unsuitable for inclusion by the investigator;
5. Have participated in an "interventional" clinical trial within the past 30 days and have taken the experimental drug;
6. Unsuitable for this trial determined by the researchers;
7. Failure to collect blood on time according to plan;
8. The blood sample does not meet the requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study aims to enroll 2430 participants from Zhongshan Hospital, Xuhui central hospitial, Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University and Shanghai Public Health Clinical Center.
Sampling Method: Non-Probability Sample
Enrollment: 2430 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Establish ctDNA-targeted sequencing models for early detection of esophageal, gastric, colorectal and hepatocellular cancer, and evaluate the diagnosis value | assessed up to 1 year
  To discover the characteristic targets of ctDNA methylation, fragment, and mutation in esophageal, gastric, colorectal cancers, and hepatocellular carcinoma, and establish the early detection panel. Then, evaluate the sensitivity and specificity of multi-cancer early detection models.
Establish and evaluate the non-invasive early detection model for hepatocellular carcinoma | assessed up to 1 year
  To establish and evaluate the early detection model for hepatocellular carcinoma based on ctDNA methylation detection, ctDNA low-pass WGS, miRNA7™ and CTC detection.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, Doctor, Study Director — Fudan University; Yunshi Zhong, Doctor, Study Director — Fudan University; Rui Liu, Doctor, Principal Investigator — Singlera Genomics Inc.; Bin Yan, Doctor, Study Director — Shanghai Zhongshan Hospital; Dongli He, Master, Study Director — Xuhui Central Hospital, Shanghai
Locations (4):
- China (4):
  - Xuhui Central Hospital, Shanghai, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Qingpu Branch of Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo S, Diep D, Plongthongkum N, Fung HL, Zhang K, Zhang K. Identification of methylation haplotype blocks aids in deconvolution of heterogeneous tissue samples and tumor tissue-of-origin mapping from plasma DNA. Nat Genet. 2017 Apr;49(4):635-642. doi: 10.1038/ng.3805. Epub 2017 Mar 6. PMID 28263317
- [Background] Chen X, Gole J, Gore A, He Q, Lu M, Min J, Yuan Z, Yang X, Jiang Y, Zhang T, Suo C, Li X, Cheng L, Zhang Z, Niu H, Li Z, Xie Z, Shi H, Zhang X, Fan M, Wang X, Yang Y, Dang J, McConnell C, Zhang J, Wang J, Yu S, Ye W, Gao Y, Zhang K, Liu R, Jin L. Non-invasive early detection of cancer four years before conventional diagnosis using a blood test. Nat Commun. 2020 Jul 21;11(1):3475. doi: 10.1038/s41467-020-17316-z. PMID 32694610
- [Derived] Huang A, Guo DZ, Su ZX, Zhong YS, Liu L, Xiong ZG, He DL, Yan B, Li QL, Feng Z, Wang WQ, Lu PX, He MJ, Qi ZP, Guo Q, Cheng JW, Zhang SY, Guo W, Li Q, Lin GY, Sun HC, Qiu SJ, He QY, Fan J, Goel A, Liu R, Jin G, Yang XR, Zhou J. GUIDE: a prospective cohort study for blood-based early detection of gastrointestinal cancers using targeted DNA methylation and fragmentomics sequencing. Mol Cancer. 2025 Jun 5;24(1):163. doi: 10.1186/s12943-025-02367-x. PMID 40468355
- [Derived] Guo DZ, Huang A, Wang YC, Zhou S, Wang H, Xing XL, Zhang SY, Cheng JW, Xie KH, Yang QC, Ma CC, Li Q, Chen Y, Su ZX, Fan J, Liu R, Liu XL, Zhou J, Yang XR. Early detection and prognosis evaluation for hepatocellular carcinoma by circulating tumour DNA methylation: A multicentre cohort study. Clin Transl Med. 2024 May;14(5):e1652. doi: 10.1002/ctm2.1652. PMID 38741204